CLINICAL TRIAL: NCT00488709
Title: FLAT: Fludarabine, Cytarabine and Topotecan in Treating Patients With Refractory or Relapsed Acute Myeloid Leukemia
Brief Title: Fludarabine, Cytarabine, Topotecan in Treating Patients With Relapsed or Refractory Acute Myeloid Leukemia
Acronym: FLAT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: PETHEMA Foundation (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LAMR 2003; FLAT
Record Dates: First submitted 2007-06-01; First posted 2007-06-20 (Estimated); Last update posted 2008-11-18 (Estimated); Status verified 2008-11

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; Multi Drug Resistance
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Topotecan; fludarabine; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Topotecan
Drug: Fludarabine
Drug: Cytarabine

SUMMARY:
The study is designed with drugs used frequently in the treatment of AML, but with a new combination less toxic,and effective in AML multidrug resistant.

Justification:

* The AML patients with primary resistance or relapsed in the first 12 months after CR, have second line chemotherapy low response rate .
* These patients with AML with primary resistance or relapse, that reach remission after a rescue treatment, have an interval free survival and a global survival very short
* Probably the resistance to the treatments is in relation to different forms expression of the MDR.
* Complete remission is considered valid evaluation, because every patient who should obtain a CR can be considered to be eligible for a possible curative treatment: Ara-C administration to high doses or the TPH treatment

DETAILED DESCRIPTION:
It is a protocol opened, multicentric, led to end to increase a) the rate of complete responses, b) the duration of the response, c) the free survival of disease and d) the global survival.

The included subjects will be patients with primary or secondary AML that they have not achieved the CR after the standard treatment with an anthracycline or derivative associated with Ara-C or have relapsed in the first 12 months after having achieved the RC. Also patients with AML that, for any reason, they could not receive the standard treatment with anthracycline and Ara-C, will be included

Cycle of induction. The patients will be treated by FLAT according to the following scheme:

* FLUDARABINE, 30 mg/m2 i.v. (In 1 hour) on the 1st to 4.
* CITARABINE, 2 g/m2 i.v. (In 4 hours), four hours after finishing the fludarabine, on the 1st to 4.
* TOPOTECAN, 1,5 mg/m2 i.v. (In 4 hours), four hours after finishing the cytarabine, on the 1st to 4.

When the patient starts recovering the hematological counts, and providing that has not blasts in the peripheral blood (SP), he will become a medullar revision (MO):

* If MO presents severe hypocellularity without blasts,no therapeutic measurement will take and there will repeat revisions weekly and MDR's study up to the CR or the blasts appearance.
* If in MO persist blasts (>5 %) but have diminished less than 50 % of the initial number, the induction will be continued by the FLAT's second shift.
* If in MO persists more than 50 % of blasts of the initial number, the patient goes out of the protocol and it will be treated as an agreement by the criterion of the center.

The patients who have managed to enter CR will receive a cycle of consolidation as soon as possible and always within 2 months from the day in which they received first FLAT's dose. The cycle of consolidation consists of another FLAT's scheme to the same doses.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects of 18 years of age or major, with diagnosis of primary or secondary AML, confirmed cytologically, that fulfill one of the following conditions:

   * Do not reach a CR after the conventional treatment.
   * Relapse in the first 12 months after a CR. During remission, patients can have be treated by a transplant. The relapse is defined as the presence of blasts in peripheric blood or the presence of >5 % of blasts in MO.
   * Not participation in a clinical trial.
2. ECOG < o = 2
3. Considered suitable patients for an intensive chemotherapy
4. Informed consent

Exclusion Criteria:

1. Pelvic or spinal radiotherapy in 4 weeks before the incorporation in the protocol.
2. Acute promyelocytic leukaemia
3. First line chemotherapy for AML which has contained fludarabine or topotecan.
4. Active or chronic hepatitis or hepatic cirrhosis.
5. Positivity known to the virus of the human immunodeficiency (HIV)
6. Pregnant or breastfeeding patients.
7. Patients with deterioration of the functions hepatic or renal, defined for the following values base them of laboratory:

   * AST or ALT >2,5 times the top limit of the normality of the center (LSNC)
   * Alkaline phosphatase >2,5 times the LSNC
   * Total bilirubin value >2 times the LSNC
   * Creatinine value >2 times the LSNC after a suitable hydration
8. Precedents of intervention of major surgery in 2 weeks before the incorporation in the protocol.
9. Patients with disease serious or not controlled (for example not controlled diabetes, infection, hypertension, etc.).
10. Patients who have received other cytotoxic drugs (except hydroxyurea to reduce the leucocytosis) as treatment of the current relapse or of the resistance, in 4 weeks before the protocol.
11. Patients with hypersensitivity known to someone of the drugs of the protocol.
12. Patients treated previously with growth factors with purposes of sensibilization.
13. Patients with psychological, intellectual or sensitive dysfunction that can reduce his capacity of comprehension and fulfillment of the protocol.
14. Patients treated before with FLAT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2003-05; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
To treat with the combination FLAT patients with acute myeloid leukaemia that they present a primary resistance | one month
•To treat with the combination FLAT a relapse in the first 12 months after reach the first CR with standard treatment | one month
To treat with combination FLAT patients can't receive the standard treatment due any cause | one month

SECONDARY OUTCOMES:
Improve the interval free survival and global survival | one year
To avoid the toxicities produced by other chemotherapy in this type of patients | 4 months
To determine the existing association between the response to the treatment with FLAT and the expression of Multi Drug Resistance (MDR) in the acute myeloid leukaemia | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Bueno Javier, Dr, Study Chair — Hospital Vall d'Hebron; Sanchez Eva, Dr, Principal Investigator — Hospital Vall d'Hebron
Locations (16):
- Spain (16):
  - Hospital Juan Canalejo, A Coruña
  - Hospital Ntra. Sra. de Sonsoles, Ávila
  - Hospital germans Trias i Pujol, Badalona
  - Centro Médico Teknon, Barcelona
  - Hospital Sant Pau, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital General Yagüe, Burgos
  - Hospital de Jerez, Cadiz
  - Complejo hospitalario Xeral-Calde, Lugo
  - Hospital Clínico Universitario San Carlos, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Hospital Virgen de la Victoria, Málaga
  - Hosptal Joan XXIII, Tarragona
  - Hospital Verge de la Cinta, Tortosa
  - Hospital Rio Hortega, Valladolid
  - Hospital Clinico Lozano Blesa, Zaragoza

REFERENCES:
- [Background] Bishop JF. The treatment of adult acute myeloid leukemia. Semin Oncol. 1997 Feb;24(1):57-69. PMID 9045305
- [Background] Stone RM. Treatment of acute myeloid leukemia: state-of-the-art and future directions. Semin Hematol. 2002 Jul;39(3 Suppl 2):4-10. doi: 10.1053/shem.2002.35977. PMID 12214287
- [Background] Lister TA, Rohatiner AZ. The treatment of acute myelogenous leukemia in adults. Semin Hematol. 1982 Jul;19(3):172-92. PMID 7051288
- [Background] Cassileth PA, Harrington DP, Appelbaum FR, Lazarus HM, Rowe JM, Paietta E, Willman C, Hurd DD, Bennett JM, Blume KG, Head DR, Wiernik PH. Chemotherapy compared with autologous or allogeneic bone marrow transplantation in the management of acute myeloid leukemia in first remission. N Engl J Med. 1998 Dec 3;339(23):1649-56. doi: 10.1056/NEJM199812033392301. PMID 9834301
- [Background] Rees JK, Gray RG, Swirsky D, Hayhoe FG. Principal results of the Medical Research Council's 8th acute myeloid leukaemia trial. Lancet. 1986 Nov 29;2(8518):1236-41. doi: 10.1016/s0140-6736(86)92674-7. PMID 2878130
- [Background] Vey N, Keating M, Giles F, Cortes J, Beran M, Estey E. Effect of complete remission on survival in patients with acute myelogenous leukemia receiving first salvage therapy. Blood. 1999 May 1;93(9):3149-50. No abstract available. PMID 10336269
- [Background] Del Poeta G, Venditti A, Aronica G, Stasi R, Cox MC, Buccisano F, Bruno A, Tamburini A, Suppo G, Simone MD, Epiceno AM, Del Moro B, Masi M, Papa G, Amadori S. P-glycoprotein expression in de novo acute myeloid leukemia. Leuk Lymphoma. 1997 Oct;27(3-4):257-74. doi: 10.3109/10428199709059682. PMID 9402325
- [Background] Germann UA. P-glycoprotein--a mediator of multidrug resistance in tumour cells. Eur J Cancer. 1996 Jun;32A(6):927-44. doi: 10.1016/0959-8049(96)00057-3. No abstract available. PMID 8763334
- [Background] Keating MJ, Kantarjian H, Smith TL, Estey E, Walters R, Andersson B, Beran M, McCredie KB, Freireich EJ. Response to salvage therapy and survival after relapse in acute myelogenous leukemia. J Clin Oncol. 1989 Aug;7(8):1071-80. doi: 10.1200/JCO.1989.7.8.1071. PMID 2666590
- [Background] Nussler V, Pelka-Fleischer R, Zwierzina H, Nerl C, Beckert B, Gieseler F, Diem H, Ledderose G, Gullis E, Sauer H, Wilmanns W. P-glycoprotein expression in patients with acute leukemia-clinical relevance. Leukemia. 1996 Jul;10 Suppl 3:S23-S31. PMID 8656697
- [Background] Hendricks CB, Rowinsky EK, Grochow LB, Donehower RC, Kaufmann SH. Effect of P-glycoprotein expression on the accumulation and cytotoxicity of topotecan (SK&F 104864), a new camptothecin analogue. Cancer Res. 1992 Apr 15;52(8):2268-78. PMID 1348448
- [Background] Michelutti A, Michieli M, Damiani D, Melli C, Ermacora A, Grimaz S, Candoni A, Russo D, Fanin R, Baccarani M. Effect of fludarabine and arabinosylcytosine on multidrug resistant cells. Haematologica. 1997 Mar-Apr;82(2):143-7. PMID 9175315
- [Background] Leoni F, Ciolli S, Nozzoli C, Santini V, Fanci R, Rossi Ferrini P. Fludarabine, cytarabine and topotecan (FLAT) as induction therapy for acute myeloid leukemia in the elderly: a preliminary report. Haematologica. 2001 Jan;86(1):104. No abstract available. PMID 11146581
- [Background] Frewin RJ, Johnson SA. The role of purine analogue combinations in the management of acute leukemias. Hematol Oncol. 2001 Dec;19(4):151-7. doi: 10.1002/hon.686. PMID 11754391
- [Background] Seiter K, Feldman EJ, Halicka HD, Traganos F, Darzynkiewicz Z, Lake D, Ahmed T. Phase I clinical and laboratory evaluation of topotecan and cytarabine in patients with acute leukemia. J Clin Oncol. 1997 Jan;15(1):44-51. doi: 10.1200/JCO.1997.15.1.44. PMID 8996123
- [Background] Sierra J, Brunet S, Granena A, Olive T, Bueno J, Ribera JM, Petit J, Besses C, Llorente A, Guardia R, Macia J, Rovira M, Badell I, Vela E, Diaz de Heredia C, Vivancos P, Carreras E, Feliu E, Montserrat E, Julia A, Cubells J, Rozman C, Domingo A, Ortega JJ. Feasibility and results of bone marrow transplantation after remission induction and intensification chemotherapy in de novo acute myeloid leukemia. Catalan Group for Bone Marrow Transplantation. J Clin Oncol. 1996 Apr;14(4):1353-63. doi: 10.1200/JCO.1996.14.4.1353. PMID 8648394
- [Background] Mayer RJ, Davis RB, Schiffer CA, Berg DT, Powell BL, Schulman P, Omura GA, Moore JO, McIntyre OR, Frei E 3rd. Intensive postremission chemotherapy in adults with acute myeloid leukemia. Cancer and Leukemia Group B. N Engl J Med. 1994 Oct 6;331(14):896-903. doi: 10.1056/NEJM199410063311402. PMID 8078551
- [Background] Bennett CL, Smith TJ, Weeks JC, Bredt AB, Feinglass J, Fetting JH, Hillner BE, Somerfield MR, Winn RJ. Use of hematopoietic colony-stimulating factors: the American Society of Clinical Oncology survey. The Health Services Research Committee of the American Society of Clinical Oncology. J Clin Oncol. 1996 Sep;14(9):2511-20. doi: 10.1200/JCO.1996.14.9.2511. PMID 8823330
- See also: Spanish association of Haematology — http://www.aehh.org